CLINICAL TRIAL: NCT03906071
Title: A Randomized Phase 3 Study of Sitravatinib in Combination With Nivolumab Versus Docetaxel in Patients With Advanced Non-Squamous Non-Small Cell Lung Cancer With Disease Progression On or After Platinum-Based Chemotherapy and Checkpoint Inhibitor Therapy SAPPHIRE
Brief Title: Phase 3 Study of Sitravatinib Plus Nivolumab vs Docetaxel in Patients With Advanced Non-Squamous Non-Small Cell Lung Cancer
Acronym: SAPPHIRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mirati Therapeutics Inc. (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA248-0001; CA248-0001 (Other: Bristol-Myers Squibb Protocol ID); 516-005 (Other: Mirati Therapeutics Protocol ID)
Record Dates: First submitted 2019-04-04; First posted 2019-04-08 (Actual); Results first posted 2024-06-25 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Non-Squamous Non-Small Cell Lung Cancer
Keywords: Sitravatinib; Nivolumab; Docetaxel; Checkpoint inhibitor; MGCD516; NSCLC; SAPPHIRE
MeSH Terms: interventions — Nivolumab; sitravatinib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nivolumab and Sitravatinib (Experimental): Nivolumab will be administered by intravenous infusion over 30 minutes at 240 mg every 2 weeks or at 480 mg every 4 weeks. Sitravatinib capsules will be administered orally, once daily.
  Interventions: Biological: Nivolumab; Drug: Sitravatinib
- Docetaxel (Active Comparator): Docetaxel will be administered by intravenous infusion at 75 mg/m2 over 1 hour every 3 weeks.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Biological: Nivolumab — Nivolumab is an antibody directed at the programmed death receptor-1 (PD-1), blocking its interaction with PD-L1 and PD-L2.
  Other Names: Opdivo
  Arms: Nivolumab and Sitravatinib
Drug: Sitravatinib — Sitravatinib is a small molecule inhibitor of receptor tyrosine kinases.
  Other Names: MGCD516
  Arms: Nivolumab and Sitravatinib
Drug: Docetaxel — Docetaxel is an anti-neoplastic agent that acts by disrupting the microtubular network in cells.
  Other Names: Taxotere
  Arms: Docetaxel

SUMMARY:
This study will compare the efficacy of the investigational agent sitravatinib in combination with nivolumab versus docetaxel in patients with advanced non-squamous NSCLC who have previously experienced disease progression on or after platinum-based chemotherapy and checkpoint inhibitor therapy.

DETAILED DESCRIPTION:
Sitravatinib (MGCD516) is an orally-available, small molecule inhibitor of a closely related spectrum of receptor tyrosine kinases (RTKs) including MET, TAM (Tyro3, AXL, MERTK) family, VEGFR family, PDGFR family, KIT, FLT3, TRK family, RET, DDR2, and selected EPH family members. Nivolumab is a human IgG monoclonal antibody that binds to the PD-1 receptor and selectively blocks the interaction with its ligands PD-L1 and PD-L2, thereby releasing PD-1 pathway mediated inhibition of the immune response, including anti-tumor immune response. RTKs have been implicated in mediating an immunosuppressive tumor microenvironment, which has emerged as a potential resistance mechanism to checkpoint inhibitor therapy. Inhibition of these RTKs by sitravatinib may augment anti-tumor immune response and improve outcomes by overcoming resistance to checkpoint inhibitor therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Non-Squamous Non-Small Cell Lung Cancer
* Receipt of at least one but not more than two prior treatment regimens in the advanced setting
* Prior treatment with PD-1/PD-L1 checkpoint inhibitor therapy and platinum-based chemotherapy in combination or in sequence (i.e., platinum-based chemotheraphy followed by checkpoint inhibitor therapy)
* Most recent treatment regimen must have included a checkpoint inhibitor therapy with radiographic disease progression on or after treatment
* Candidate to receive docetaxel as second or third line therapy

Exclusion Criteria:

* Uncontrolled brain metastases
* Tumors that have tested positive for EGFR, ROS1, ALK mutations, or ALK fusions
* Unacceptable toxicity with prior checkpoint inhibitor therapy
* Receipt of systemic anti-cancer therapy post checkpoint inhibitor therapy, other than maintenance chemotherapy
* Impaired heart function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 577 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2025-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (261):
- United States (133):
  - Local Institution - 005-164, Birmingham, Alabama
  - Clearview Cancer Institute - Huntsville, Huntsville, Alabama
  - Palo Verde Cancer Specialists - Glendale, Glendale, Arizona
  - The Oncology Institute of Hope & Innovation - Tucson, Tucson, Arizona
  - Yuma Regional Medical Center, Yuma, Arizona
  - Local Institution - 005-174, Jonesboro, Arkansas
  - NEA Baptist Fowler Family Center for Cancer Care, Jonesboro, Arkansas
  - Highlands Oncology Group - Springdale, Springdale, Arkansas
  - Comprehensive Blood and Cancer Center - Bakersfield, Bakersfield, California
  - Local Institution - 005-118, Beverly Hills, California
  - Local Institution - 005-171, Fresno, California
  - Providence Medical Foundation - Virginia K. Crosson Cancer Center - Fullerton, Fullerton, California
  - Local Institution - 005-096, Long Beach, California
  - Cancer and Blood Specialty Clinic, Los Alamitos, California
  - Los Angeles Hematology Oncology Medical Group, Los Angeles, California
  - Local Institution - 005-185, Los Angeles, California
  - Local Institution - 005-072, Newport Beach, California
  - Local Institution - 005-109, Northridge, California
  - Local Institution - 005-177, Redlands, California
  - Local Institution - 005-112, Riverside, California
  - University of California San Francisco, San Francisco, California
  - Local Institution - 005-176, San Marcos, California
  - Local Institution - 005-192, Torrance, California
  - Local Institution - 005-090, West Covina, California
  - Local Institution - 005-105, Whittier, California
  - Local Institution - 005-097, Lafayette, Colorado
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Michael and Dianne Bienes Comprehensive Cancer Center, Fort Lauderdale, Florida
  - Local Institution - 005-120, Fort Myers, Florida
  - Memorial Regional Hospital, Hollywood, Florida
  - Watson Clinic Cancer and Research Center, Lakeland, Florida
  - Mount Sinai Health System, Miami Beach, Florida
  - Local Institution - 005-120E, Naples, Florida
  - Local Institution - 005-079, Ocala, Florida
  - Local Institution - 005-104, Orlando, Florida
  - SCRI - Florida Cancer Specialists - North Region Research Office, St. Petersburg, Florida
  - SCRI - Florida Cancer Specialists - Panhandle Research Office, Tallahassee, Florida
  - Local Institution - 005-154, West Palm Beach, Florida
  - University Cancer & Blood Center (UCBC) - Athens, Athens, Georgia
  - Local Institution - 005-146, Atlanta, Georgia
  - John B. Amos Cancer Center Research, Columbus, Georgia
  - Local Institution - 005-119, Marietta, Georgia
  - Straub Medical Center, Honolulu, Hawaii
  - Local Institution - 005-191, Coeur d'Alene, Idaho
  - Local Institution - 005-151, Chicago, Illinois
  - Local Institution - 005-110, Evanston, Illinois
  - Local Institution - 005-198, Niles, Illinois
  - Orchard Healthcare Research, Skokie, Illinois
  - Healthcare Research Network - Tinley Park, Tinley Park, Illinois
  - Fort Wayne Medical Oncology and Hematology - Fort Wayne South Office, Fort Wayne, Indiana
  - Local Institution - 005-122, Goshen, Indiana
  - Franciscan Health Cancer Center Indianapolis, Indianapolis, Indiana
  - Local Institution - 005-150, Lafayette, Indiana
  - Local Institution - 005-169, Westwood, Kansas
  - Local Institution - 005-098, Wichita, Kansas
  - Commonwealth Cancer Center - Frankfort, Danville, Kentucky
  - Local Institution - 005-153, Louisville, Kentucky
  - New England Cancer Specialists - Scarborough, Scarborough, Maine
  - Local Institution - 005-178, Rockville, Maryland
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Local Institution - 005-127, Minneapolis, Minnesota
  - Local Institution - 005-159, Saint Louis Park, Minnesota
  - Jackson Oncology Associates - The Hederman Cancer Center, Jackson, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Kansas City Care Health Center - Research Medical Campus, Kansas City, Missouri
  - Sisters of Charity of Leavenworth Health St. Marys, Billings, Montana
  - Saint Francis Cancer Treatment Center, Grand Island, Nebraska
  - Methodist Hospital - Omaha, Omaha, Nebraska
  - The Oncology Institute of Hope & Innovation - Henderson, Henderson, Nevada
  - Local Institution - 005-152, Henderson, Nevada
  - Local Institution - 005-142, Florham Park, New Jersey
  - Local Institution - 005-163, Little Silver, New Jersey
  - Cooperman Barnabas Medical Center, Livingston, New Jersey
  - Regional Cancer Care Associates - Sparta, Sparta, New Jersey
  - Local Institution - 005-123, Johnson City, New York
  - Local Institution - 005-182, Lake Success, New York
  - New York Cancer & Blood Specialists - Port Jefferson Medical Oncology, Port Jefferson Station, New York
  - Local Institution - 005-107, Stony Brook, New York
  - Local Institution - 005-196, Canton, Ohio
  - USOR - Oncology Hematology Care - Blue Ash, Cincinnati, Ohio
  - Local Institution - 005-181, Columbus, Ohio
  - Tricounty Hematology and Oncology - Massillon, Massillon, Ohio
  - Local Institution - 005-103, Toledo, Ohio
  - Local Institution - 005-088, Oklahoma City, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - Local Institution - 005-073, Portland, Oregon
  - USOR - Alliance Cancer Specialists - Horsham (Abington Hematology Oncology Associates), Horsham, Pennsylvania
  - Local Institution - 005-186, Philadelphia, Pennsylvania
  - Local Institution - 005-137A, Dickson, Tennessee
  - Local Institution - 005-137B, Dickson, Tennessee
  - Local Institution - 005-137C, Dickson, Tennessee
  - Local Institution - 005-137D, Dickson, Tennessee
  - Local Institution - 005-137E, Dickson, Tennessee
  - Local Institution - 005-137F, Dickson, Tennessee
  - Local Institution - 005-137G, Dickson, Tennessee
  - Local Institution - 005-137H, Dickson, Tennessee
  - Local Institution - 005-137I, Dickson, Tennessee
  - Local Institution - 005-137J, Dickson, Tennessee
  - Local Institution - 005-137K, Dickson, Tennessee
  - Local Institution - 005-137L, Dickson, Tennessee
  - Local Institution - 005-137M, Hendersonville, Tennessee
  - Local Institution - 005-195, Memphis, Tennessee
  - Local Institution - 005-137, Nashville, Tennessee
  - Local Institution - 005-134, Austin, Texas
  - Local Institution - 005-075, Beaumont, Texas
  - Local Institution - 005-128, Dallas, Texas
  - Local Institution - 005-129, Dallas, Texas
  - Local Institution - 005-126, Dallas, Texas
  - USOR - Texas Oncology Northeast Texas - Denison, Denison, Texas
  - Local Institution - 005-124, Denton, Texas
  - The Center for Cancer & Blood Disorders - Fort Worth, Fort Worth, Texas
  - Oncology Consultants - Texas Medical Center, Houston, Texas
  - Local Institution - 005-076, Houston, Texas
  - Millennium Research and Clinical Development, Houston, Texas
  - USOR - US Oncology Investigational Products Center, Irving, Texas
  - Local Institution - 005-125, McKinney, Texas
  - Texas Oncology - San Antonio Medical Center, San Antonio, Texas
  - USOR - Texas Oncology - Sugar Land, Sugar Land, Texas
  - USOR - Texas Oncology Northeast Texas - Cancer and Research Institute - Tyler, Tyler, Texas
  - Local Institution - 005-144, Charlottesville, Virginia
  - Hematology Oncology Associates of Fredericksburg, Fredericksburg, Virginia
  - Virginia Cancer Institute - West End, Richmond, Virginia
  - Overlake Medical Center and Clinics, Bellevue, Washington
  - Local Institution - 005-082, Everett, Washington
  - Local Institution - 005-111, Seattle, Washington
  - Local Institution - 005-187, Spokane, Washington
  - Local Institution - 005-081, Tacoma, Washington
  - Northwest Medical Specialties - Tacoma, Tacoma, Washington
  - Local Institution - 005-136, Vancouver, Washington
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Local Institution - 005-116, Madison, Wisconsin
  - Froedtert Hospital, Milwaukee, Wisconsin
- Belgium (8):
  - Local Institution - 005-201, Brasschaat
  - Local Institution - 005-200, Charleroi
  - Local Institution - 005-206, Edegem
  - Local Institution - 005-202, Ghent
  - Local Institution - 005-207, Ghent
  - Local Institution - 005-205, Roeselare
  - Local Institution - 005-204, Ronse
  - Centre Hospitalier Universitaire Universite Catholique de Louvain - Site Godinne, Yvoir
- Canada (9):
  - Local Institution - 005-259, Calgary, Alberta
  - Local Institution - 005-250, Moncton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Local Institution - 005-252, Hamilton, Ontario
  - Local Institution - 005-251, Toronto, Ontario
  - Local Institution - 005-257, Windsor, Ontario
  - Local Institution - 005-255, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - Local Institution - 005-258, Québec
- France (16):
  - Local Institution - 005-307, Brest
  - Local Institution - 005-310, Bron
  - Local Institution - 005-311, Créteil
  - Local Institution - 005-303, Dijon
  - Local Institution - 005-309, Le Mans
  - Local Institution - 005-308, Limoges
  - Local Institution - 005-317, Lyon
  - Local Institution - 005-301, Marseille
  - Local Institution - 005-312, Marseille
  - Local Institution - 005-313, Montpellier
  - Local Institution - 005-306, Mulhouse
  - Local Institution - 005-302, Paris
  - Local Institution - 005-314, Rouen
  - Local Institution - 005-316, Saint-Herblain
  - Local Institution - 005-305, Strasbourg
  - Local Institution - 005-304, Villejuif
- Germany (16):
  - Local Institution - 005-400, Bad Berka
  - Local Institution - 005-418, Berlin
  - Local Institution - 005-401, Bonn
  - Local Institution - 005-412, Cologne
  - Local Institution - 005-419, Essen
  - Local Institution - 005-406, Esslingen am Neckar
  - Local Institution - 005-403, Gauting
  - Local Institution - 005-417, Grohansdorf
  - Local Institution - 005-408, Halle
  - Local Institution - 005-411, Immenstadt im Allgäu
  - Local Institution - 005-416, Kassel
  - Local Institution - 005-410, Löwenstein
  - Local Institution - 005-405, Lübeck
  - Local Institution - 005-414, Mainz
  - Local Institution - 005-413, München
  - Local Institution - 005-402, München
- Hungary (8):
  - Local Institution - 005-454, Budapest
  - Local Institution - 005-457, Budapest
  - Local Institution - 005-455, Budapest
  - Local Institution - 005-453, Farkasgyepű
  - Local Institution - 005-452, Győr
  - Local Institution - 005-451, Szombathely
  - Local Institution - 005-450, Tatabánya
  - Local Institution - 005-456, Törökbálint
- Israel (7):
  - Local Institution - 005-500, Afula
  - Local Institution - 005-501, Beer Yaakov
  - Local Institution - 005-504, Beersheba
  - Local Institution - 005-502, Holon
  - Local Institution - 005-507, Jerusalem
  - Local Institution - 005-506, Ramat Gan
  - Local Institution - 005-505, Zsfat
- Italy (14):
  - Local Institution - 005-612, Alessandria
  - Local Institution - 005-602, Bari
  - Local Institution - 005-603, Catania
  - Local Institution - 005-611, Cremona
  - Local Institution - 005-608, Lecce
  - Local Institution - 005-610, Meldola
  - Local Institution - 005-606, Milan
  - Local Institution - 005-605, Monza
  - Local Institution - 005-604, Napoli
  - Local Institution - 005-600, Parma
  - Local Institution - 005-607, Piacenza
  - Local Institution - 005-609, Pisa
  - Local Institution - 005-614, Roma
  - Ospedale di Circolo e Fondazione Macchi, Varese
- Netherlands (14):
  - Local Institution - 005-700, 's-Hertogenbosch
  - Local Institution - 005-703, Amsterdam
  - Local Institution - 005-711, Amsterdam
  - Local Institution - 005-707, Breda
  - Local Institution - 005-713, Dordrecht
  - Local Institution - 005-702, Groningen
  - Local Institution - 005-712, Maastricht
  - Local Institution - 005-714, Nijmegen
  - Local Institution - 005-710, Rotterdam
  - Local Institution - 005-705, Rotterdam
  - Local Institution - 005-709, The Hague
  - Local Institution - 005-701, Utrecht
  - Local Institution - 005-708, Utrecht
  - Local Institution - 005-706, Zwolle
- Spain (24):
  - Local Institution - 005-807, A Coruña
  - Local Institution - 005-800, Badalona
  - Local Institution - 005-822, Barcelona
  - Local Institution - 005-811, Barcelona
  - Local Institution - 005-810, Barcelona
  - Local Institution - 005-805, Jaén
  - Local Institution - 005-816, Las Palmas de Gran Canaria
  - Local Institution - 005-817, León
  - Local Institution - 005-812, Lugo
  - Hospital Universitario La Princesa, Madrid
  - Local Institution - 005-808, Madrid
  - Local Institution - 005-819, Madrid
  - Local Institution - 005-821, Madrid
  - Local Institution - 005-813, Madrid
  - Local Institution - 005-815, Madrid
  - Local Institution - 005-809, Madrid
  - Hospital Universitario La Paz, Madrid
  - Local Institution - 005-806, Majadahonda
  - Local Institution - 005-801, Málaga
  - Local Institution - 005-803, Oviedo
  - Local Institution - 005-823, Santiago de Compostela
  - IVO - Fundacion Instituto Valenciano de Oncologia, Valencia
  - Local Institution - 005-804, Valencia
  - Local Institution - 005-818, Vigo
- Switzerland (4):
  - Inselspital Universitatsspital Bern, Bern
  - Hopitaux Universitaires de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois Lausanne, Lausanne
  - Kantonsspital Winterthur, Winterthur
- United Kingdom (8):
  - Velindre University NHS Trust, Cardiff
  - Local Institution - 005-904, Cornwall
  - University Hospitals of Leicester NHS Trust, Leicester
  - Local Institution - 005-908, London
  - Local Institution - 005-900, London
  - The Royal Marsden NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - Local Institution - 005-903, Middlesex

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Nivolumab and Sitravatinib: Participants with Advanced Non-Squamous Non-Small Cell Lung Cancer were administered with Nivolumab by intravenous infusion over 30 minutes at 240 milligram (mg) every 2 weeks or at 480 mg every 4 weeks at the discretion of the investigator . Sitravatinib capsules were administered at 100 mg orally, once daily.
- Docetaxel: Participants with Advanced Non-Squamous Non-Small Cell Lung Cancer were administered with Docetaxel by intravenous infusion at 75 milligram per meter square (mg/m^2) over 1 hour every 3 weeks.
Period: Overall Study
Arm/Group | Nivolumab and Sitravatinib | Docetaxel
Started (The intent-to-treat (ITT) population is defined as all patients who are randomized into this study.) | 284 | 293
Safety Population (The Safety Population is defined as all patients who received any dose of study medication (i.e., sitravatinib, nivolumab or docetaxel).) | 281 | 273
Completed (Continuing in the study.) | 84 | 77
Not Completed | 200 | 216
Not completed — Death | 180 | 185
Not completed — Lost to Follow-up | 3 | 3
Not completed — Withdrawal by Subject | 15 | 27
Not completed — Other | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab and Sitravatinib | Docetaxel | Total
Number analyzed (Participants) | 284 | 293 | 577
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (8.48) | 65.0 (10.08) | 65.0 (9.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 125 | 239
  Male | 170 | 168 | 338
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 18 | 30
  Not Hispanic or Latino | 219 | 207 | 426
  Unknown or Not Reported | 53 | 68 | 121
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 7 | 9 | 16
  Black or African American | 8 | 14 | 22
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  White | 211 | 198 | 409
  Other | 4 | 3 | 7
  Not Reported | 34 | 46 | 80
  Unknown | 5 | 4 | 9
  Missing | 14 | 18 | 32

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS is defined as time from date of randomization to date of death due to any cause. Patients who did not die on study are censored at the date of the last on-study follow-up that the patient was known to be alive (including follow-up data). Results obtained via Kaplan-Meier estimation, Brookmeyer and Crowley (1982) method.
Time Frame: From randomization date to date of death due to any cause (Up to approximately 44 months)
Population: Intent-to-Treat population: all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab and Sitravatinib | Docetaxel
Number analyzed (Participants) | 284 | 293
Months | 12.22 [10.41 to 13.93] | 10.58 [9.40 to 12.29]
Statistical Analysis 1: Comparison: Nivolumab and Sitravatinib vs Docetaxel; Test type: Superiority; p = 0.144, Log Rank — The p-value is based on a unstratified log-rank test. (2-Sided); Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.70 to 1.05] — Based on the unstratified cox proportional hazards model

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Event (TEAEs)
Description: An adverse event (AE) is any reaction, side effect or other undesirable medical event that occurs during participation in a clinical trial, regardless of treatment group or suspected causal relationship to study treatment. Serious adverse events (SAE) are defined as any AE which results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; constitutes an important medical event. A treatment emergent AE (TEAE) is an AE that occurs after the first dose of any study treatment or any preexisting condition that increases in severity after the first dose of study treatment. Adverse events were graded using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 (Grade 3 = Severe, Grade 4 = Life-threatening, Grade 5 = Death).
Time Frame: From first dose up to 28 days post last dose, and up to 100 days post last dose of nivolumab for immune-related AEs (Up to maximum of 38 months)
Population: Safety Population: all patients who received any dose of study medication (i.e., sitravatinib, nivolumab or docetaxel)
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab and Sitravatinib | Docetaxel
Number analyzed (Participants) | 281 | 273
Participants
  Any TEAE | 280 | 272
  Grade 3 or Greater TEAEs | 214 | 216
  Serious TEAEs | 126 | 101
  TEAEs Leading to Study Drug Dose Reduction or Interruption | 213 | 136
  Treatment-Related TEAEs Leading to Study Drug Dose Reduction or Interruption | 184 | 110
  Treatment-Related TEAEs Leading to Study Drug Discontinuation | 52 | 32
  TEAEs Leading to Study Discontinuation | 11 | 18
  Immune-Related TEAE | 129 | 0
  TEAE with Outcome of Death | 46 | 17
  Treatment-Related TEAEs with Outcome of Death | 1 | 3

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAE) Leading to Study Drug Discontinuation
Description: An adverse event (AE) is any reaction, side effect or other undesirable medical event that occurs during participation in a clinical trial, regardless of treatment group or suspected causal relationship to study treatment. A treatment emergent AE (TEAE) is an AE that occurs after the first dose of any study treatment or any preexisting condition that increases in severity after the first dose of study treatment.
Time Frame: as for outcome 2
Population: Safety Population: all patients who received any dose of study medication (i.e., sitravatinib, nivolumab or docetaxel)
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab and Sitravatinib | Docetaxel
Number analyzed (Participants) | 281 | 273
Participants
  Discontinuation of Study Drug | 77 | 44
  Discontinuation of Nivolumab: number analyzed (Participants) | 281 | 0
  Discontinuation of Nivolumab | 50 |
  Discontinuation of Sitravatinib: number analyzed (Participants) | 281 | 0
  Discontinuation of Sitravatinib | 74 |

4. Secondary Outcome: Number of Participants With Maximum Post Baseline Hematology Grade Results
Description: The severity of hematology results were graded based upon the participants symptoms according to the Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0); Hematology parameters were evaluated for severity according to the following scale: Grade 1 = Mild - transient or mild discomfort; no medical intervention required; Grade 2 = Moderate - mild to moderate limitation in activity; Grade 3 = Severe; Grade 4 = Life threatening; Grade 5 = Death. Number of participants with maximum post baseline grades is presented. Grade 0 is defined as absence of an AE or within normal limits. Baseline is defined as the last pre-dose assessment.
Time Frame: From first dose up to 28 days post last dose (Up to an average of 7.5 months and maximum of 36 months)
Population: Safety Population (all patients who received any dose of study medication) with at least 1 post-baseline result
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab and Sitravatinib | Docetaxel
Number analyzed (Participants) | 274 | 269
Participants
  Hemoglobin (g/L) - Anemia: Grade 0 | 118 | 27
  Hemoglobin (g/L) - Anemia: Grade 1 | 134 | 146
  Hemoglobin (g/L) - Anemia: Grade 2 | 16 | 80
  Hemoglobin (g/L) - Anemia: Grade 3 | 6 | 16
  Hemoglobin (g/L) - Anemia: Grade 4 | 0 | 0
  Hemoglobin (g/L) - Anemia: Grade 5 | 0 | 0
  Hemoglobin (g/L) increased: Grade 0 | 236 | 268
  Hemoglobin (g/L) increased: Grade 1 | 35 | 1
  Hemoglobin (g/L) increased: Grade 2 | 2 | 0
  Hemoglobin (g/L) increased: Grade 3 | 1 | 0
  Hemoglobin (g/L) increased: Grade 4 | 0 | 0
  Hemoglobin (g/L) increased: Grade 5 | 0 | 0
  Neutrophils (10^9/L) count decreased: number analyzed (Participants) | 274 | 266
  Neutrophils (10^9/L) count decreased: Grade 0 | 265 | 66
  Neutrophils (10^9/L) count decreased: Grade 1 | 8 | 7
  Neutrophils (10^9/L) count decreased: Grade 2 | 1 | 25
  Neutrophils (10^9/L) count decreased: Grade 3 | 0 | 42
  Neutrophils (10^9/L) count decreased: Grade 4 | 0 | 126
  Neutrophils (10^9/L) count decreased: Grade 5 | 0 | 0
  Platelets (10^9/L) count decreased: number analyzed (Participants) | 274 | 268
  Platelets (10^9/L) count decreased: Grade 0 | 207 | 221
  Platelets (10^9/L) count decreased: Grade 1 | 63 | 43
  Platelets (10^9/L) count decreased: Grade 2 | 3 | 3
  Platelets (10^9/L) count decreased: Grade 3 | 0 | 1
  Platelets (10^9/L) count decreased: Grade 4 | 1 | 0
  Platelets (10^9/L) count decreased: Grade 5 | 0 | 0
  Lymphocytes (10^9/L) count decreased: number analyzed (Participants) | 274 | 264
  Lymphocytes (10^9/L) count decreased: Grade 0 | 117 | 59
  Lymphocytes (10^9/L) count decreased: Grade 1 | 58 | 39
  Lymphocytes (10^9/L) count decreased: Grade 2 | 66 | 83
  Lymphocytes (10^9/L) count decreased: Grade 3 | 33 | 72
  Lymphocytes (10^9/L) count decreased: Grade 4 | 0 | 11
  Lymphocytes (10^9/L) count decreased: Grade 5 | 0 | 0
  Lymphocytes (10^9/L) count increased: number analyzed (Participants) | 274 | 264
  Lymphocytes (10^9/L) count increased: Grade 0 | 266 | 257
  Lymphocytes (10^9/L) count increased: Grade 1 | 0 | 0
  Lymphocytes (10^9/L) count increased: Grade 2 | 8 | 7
  Lymphocytes (10^9/L) count increased: Grade 3 | 0 | 0
  Lymphocytes (10^9/L) count increased: Grade 4 | 0 | 0
  Lymphocytes (10^9/L) count increased: Grade 5 | 0 | 0

5. Secondary Outcome: Number of Participants With Maximum Post Baseline Chemistry Grade Results
Description: The severity of chemistry results were graded based upon the participants symptoms according to the Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0); Chemistry parameters were evaluated for severity according to the following scale: Grade 1 = Mild - transient or mild discomfort; no medical intervention required; Grade 2 = Moderate - mild to moderate limitation in activity; Grade 3 = Severe; Grade 4 = Life threatening; Grade 5 = Death. Number of participants with maximum post baseline grades is presented. Grade 0 is defined as absence of an AE or within normal limits. Baseline is defined as the last pre-dose assessment.
Time Frame: From first dose up to 28 days post last dose (Up to an average of 7.5 months and maximum of 36 months)
Population: Safety Population (all patients who received any dose of study medication) with at least 1 post-baseline result
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab and Sitravatinib | Docetaxel
Number analyzed (Participants) | 274 | 268
Participants
  Alanine Aminotransferase (U/L) increased: number analyzed (Participants) | 274 | 266
  Alanine Aminotransferase (U/L) increased: Grade 0 | 106 | 228
  Alanine Aminotransferase (U/L) increased: Grade 1 | 151 | 37
  Alanine Aminotransferase (U/L) increased: Grade 2 | 10 | 0
  Alanine Aminotransferase (U/L) increased: Grade 3 | 7 | 1
  Alanine Aminotransferase (U/L) increased: Grade 4 | 0 | 0
  Alanine Aminotransferase (U/L) increased: Grade 5 | 0 | 0
  Aspartate Aminotransferase (U/L) increased: number analyzed (Participants) | 274 | 267
  Aspartate Aminotransferase (U/L) increased: Grade 0 | 100 | 216
  Aspartate Aminotransferase (U/L) increased: Grade 1 | 163 | 49
  Aspartate Aminotransferase (U/L) increased: Grade 2 | 8 | 2
  Aspartate Aminotransferase (U/L) increased: Grade 3 | 3 | 0
  Aspartate Aminotransferase (U/L) increased: Grade 4 | 0 | 0
  Aspartate Aminotransferase (U/L) increased: Grade 5 | 0 | 0
  Creatinine (umol/L) increased: Grade 0 | 180 | 194
  Creatinine (umol/L) increased: Grade 1 | 67 | 55
  Creatinine (umol/L) increased: Grade 2 | 27 | 19
  Creatinine (umol/L) increased: Grade 3 | 0 | 0
  Creatinine (umol/L) increased: Grade 4 | 0 | 0
  Creatinine (umol/L) increased: Grade 5 | 0 | 0
  Bilirubin (umol/L) increased: number analyzed (Participants) | 274 | 267
  Bilirubin (umol/L) increased: Grade 0 | 252 | 240
  Bilirubin (umol/L) increased: Grade 1 | 17 | 20
  Bilirubin (umol/L) increased: Grade 2 | 4 | 6
  Bilirubin (umol/L) increased: Grade 3 | 1 | 1
  Bilirubin (umol/L) increased: Grade 4 | 0 | 0
  Bilirubin (umol/L) increased: Grade 5 | 0 | 0
  Sodium (mmol/L) - Hyponatremia: Grade 0 | 147 | 147
  Sodium (mmol/L) - Hyponatremia: Grade 1 | 105 | 100
  Sodium (mmol/L) - Hyponatremia: Grade 2 | 11 | 19
  Sodium (mmol/L) - Hyponatremia: Grade 3 | 9 | 2
  Sodium (mmol/L) - Hyponatremia: Grade 4 | 2 | 0
  Sodium (mmol/L) - Hyponatremia: Grade 5 | 0 | 0
  Sodium (mmol/L) - Hypernatremia: Grade 0 | 268 | 259
  Sodium (mmol/L) - Hypernatremia: Grade 1 | 5 | 9
  Sodium (mmol/L) - Hypernatremia: Grade 2 | 0 | 0
  Sodium (mmol/L) - Hypernatremia: Grade 3 | 1 | 0
  Sodium (mmol/L) - Hypernatremia: Grade 4 | 0 | 0
  Sodium (mmol/L) - Hypernatremia: Grade 5 | 0 | 0
  Potassium (mmol/L) - Hypokalemia: Grade 0 | 217 | 222
  Potassium (mmol/L) - Hypokalemia: Grade 1 | 41 | 37
  Potassium (mmol/L) - Hypokalemia: Grade 2 | 0 | 0
  Potassium (mmol/L) - Hypokalemia: Grade 3 | 15 | 9
  Potassium (mmol/L) - Hypokalemia: Grade 4 | 1 | 0
  Potassium (mmol/L) - Hypokalemia: Grade 5 | 0 | 0
  Potassium (mmol/L) - Hyperkalemia: Grade 0 | 217 | 213
  Potassium (mmol/L) - Hyperkalemia: Grade 1 | 34 | 40
  Potassium (mmol/L) - Hyperkalemia: Grade 2 | 20 | 12
  Potassium (mmol/L) - Hyperkalemia: Grade 3 | 2 | 3
  Potassium (mmol/L) - Hyperkalemia: Grade 4 | 1 | 0
  Potassium (mmol/L) - Hyperkalemia: Grade 5 | 0 | 0
  Urate (umol/L) - Hyperuricemia: number analyzed (Participants) | 273 | 266
  Urate (umol/L) - Hyperuricemia: Grade 0 | 189 | 224
  Urate (umol/L) - Hyperuricemia: Grade 1 | 84 | 42
  Urate (umol/L) - Hyperuricemia: Grade 2 | 0 | 0
  Urate (umol/L) - Hyperuricemia: Grade 3 | 0 | 0
  Urate (umol/L) - Hyperuricemia: Grade 4 | 0 | 0
  Urate (umol/L) - Hyperuricemia: Grade 5 | 0 | 0
  Lipase (U/L) increased: number analyzed (Participants) | 273 | 263
  Lipase (U/L) increased: Grade 0 | 181 | 213
  Lipase (U/L) increased: Grade 1 | 41 | 24
  Lipase (U/L) increased: Grade 2 | 22 | 14
  Lipase (U/L) increased: Grade 3 | 20 | 9
  Lipase (U/L) increased: Grade 4 | 9 | 3
  Lipase (U/L) increased: Grade 5 | 0 | 0
  Amylase (U/L) increased: number analyzed (Participants) | 266 | 256
  Amylase (U/L) increased: Grade 0 | 184 | 213
  Amylase (U/L) increased: Grade 1 | 46 | 26
  Amylase (U/L) increased: Grade 2 | 20 | 12
  Amylase (U/L) increased: Grade 3 | 13 | 3
  Amylase (U/L) increased: Grade 4 | 3 | 2
  Amylase (U/L) increased: Grade 5 | 0 | 0
  Alkaline Phosphatase (U/L) increased: number analyzed (Participants) | 274 | 266
  Alkaline Phosphatase (U/L) increased: Grade 0 | 162 | 201
  Alkaline Phosphatase (U/L) increased: Grade 1 | 105 | 62
  Alkaline Phosphatase (U/L) increased: Grade 2 | 2 | 2
  Alkaline Phosphatase (U/L) increased: Grade 3 | 5 | 1
  Alkaline Phosphatase (U/L) increased: Grade 4 | 0 | 0
  Alkaline Phosphatase (U/L) increased: Grade 5 | 0 | 0
  Albumin (g/L) - Hypoalbuminemia: number analyzed (Participants) | 274 | 267
  Albumin (g/L) - Hypoalbuminemia: Grade 0 | 108 | 109
  Albumin (g/L) - Hypoalbuminemia: Grade 1 | 81 | 83
  Albumin (g/L) - Hypoalbuminemia: Grade 2 | 79 | 72
  Albumin (g/L) - Hypoalbuminemia: Grade 3 | 6 | 3
  Albumin (g/L) - Hypoalbuminemia: Grade 4 | 0 | 0
  Albumin (g/L) - Hypoalbuminemia: Grade 5 | 0 | 0

6. Secondary Outcome: Objective Response Rate (ORR) Per Central Radiographic Assessment
Description: ORR is defined as percentage of participants with confirmed complete response (CR) or partial response (PR) per RECIST version 1.1 recorded from randomization until disease progression or start of new anti-cancer therapy. Patients who cannot be assessed for response are counted as non-responders. CR is defined as complete disappearance of all target lesions with the exception of nodal disease; PR is defined as >=30% decrease under baseline of the sum of diameters of all target measurable lesions.
Time Frame: From randomization until disease progression or start of new anti-cancer therapy (Up to approximately 44 months)
Population: The Modified Intent-to-Treat Population: all patients who are randomized into this study and have measurable disease (per RECIST 1.1) at baseline per central radiographic assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab and Sitravatinib | Docetaxel
Number analyzed (Participants) | 282 | 290
Percentage of participants | 15.6 [11.57 to 20.37] | 17.2 [13.08 to 22.09]

7. Secondary Outcome: Duration of Response (DOR) Per Central Radiographic Assessment
Description: DOR is defined as the time from date of the first documentation of confirmed objective response (CR or PR) to the first documentation of disease progression (PD) or to death due to any cause in the absence of documented PD. Complete response (CR) is defined as complete disappearance of all target lesions with the exception of nodal disease. Partial response (PR) is defined as >=30% decrease under baseline of the sum of diameters of all target measurable lesions. Progressive Disease (PD) is defined as a 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum is observed during therapy) with a minimum absolute increase of 5 mm, or unequivocal progression of pre-existing non-target lesions. Results obtained via Kaplan-Meier estimation, Brookmeyer and Crowley (1982) method.
Time Frame: From randomization to the first documentation of disease progression (PD) or to death due to any cause in the absence of documented PD (Up to approximately 44 months)
Population: Modified Intent-to-Treat Population (all patients who are randomized into this study and have measurable disease (per RECIST 1.1) at baseline) with a confirmed objective response (CR or PR) per central radiographic assessment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab and Sitravatinib | Docetaxel
Number analyzed (Participants) | 44 | 50
Months | 7.43 [5.36 to 13.08] | 7.10 [5.85 to 11.79]

8. Secondary Outcome: Clinical Benefit Rate Per Central Radiographic Assessment
Description: CBR is defined as the percentage of patients documented to have a confirmed CR, confirmed PR, or SD, according to RECIST 1.1 as the best response. Complete response (CR) is defined as complete disappearance of all target lesions with the exception of nodal disease. Partial response (PR) is defined as >=30% decrease under baseline of the sum of diameters of all target measurable lesions. Stable Disease (SD) is concluded when the response does not qualify for CR, PR or Progression. Progression is defined as 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum is observed during therapy) with a minimum absolute increase of 5 mm.
Time Frame: From randomization until disease progression or start of new anti-cancer therapy (Up to approximately 44 months)
Population: The Modified Intent-to-Treat Population: all patients who are randomized into this study and have measurable disease (per RECIST 1.1) at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab and Sitravatinib | Docetaxel
Number analyzed (Participants) | 282 | 290
Percentage of participants | 75.5 [70.08 to 80.43] | 64.5 [58.68 to 69.99]

9. Secondary Outcome: Progression-Free Survival (PFS) Per Central Radiographic Assessment
Description: PFS is defined as the time from randomization to the date of the first documentation of objective disease progression or death due to any cause. Progressive Disease (PD) is defined as a 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum is observed during therapy) with a minimum absolute increase of 5 mm, or unequivocal progression of pre-existing non-target lesions. Censoring was assigned on the date of the last tumor assessment if no assessment of tumor progression is identified and the patient does not die while on study. Patients with no evaluation of disease after first study treatment will have PFS censored on the date of randomization. Patients who start new anti-cancer therapy prior to documented PD will be censored at the date of the last tumor assessment prior to the start of the new therapy. Results obtained using Kaplan-Meier estimation, Brookmeyer and Crowley (1982) method.
Time Frame: From randomization to the date of the first documentation of objective disease progression or death due to any cause (Up to approximately 44 months)
Population: Intent-to-Treat population: all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab and Sitravatinib | Docetaxel
Number analyzed (Participants) | 284 | 293
Months | 4.40 [3.91 to 5.42] | 5.42 [3.91 to 5.75]

10. Secondary Outcome: 1-Year Survival Rate
Description: 1-Year Survival will be defined as the percentage of participants surviving at 1 year after the first dose. Results obtained via Kaplan-Meier estimation, Greenwood's formula (1980).
Time Frame: At 12 months from first dose
Population: Intent-to-Treat Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab and Sitravatinib | Docetaxel
Number analyzed (Participants) | 284 | 293
Percentage of participants | 50.18 [44.05 to 55.99] | 44.12 [38.01 to 50.05]

11. Secondary Outcome: Change From Baseline in the Lung Cancer Symptom Scale (LCSS) Average Total Score
Description: The LCSS is a lung cancer specific measure of quality of life and includes 9 questions, including patient-reported ratings of six symptoms (appetite loss, fatigue, cough, dyspnea, hemoptysis, pain) and three summary items (symptom distress, activity level, overall quality of life) using 100-mm visual analogue scales ranging from 0 (lowest rating) to 100 (highest rating). The average total score = is a sum of items 1 to 9 divided by the total number of items (sum of items 1 to 9) / 9).
Time Frame: Clinic visit closest to the disease evaluation on weeks 9, 17, 25, 33, 41, 49.
Population: Intent-to-Treat population (all randomized participants) with available scores for each assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Nivolumab and Sitravatinib | Docetaxel
Number analyzed (Participants) | 177 | 142
Score on a scale
  Assessment 1 (Week 9) | 4.10 [1.87 to 6.33] | 2.75 [0.27 to 5.24]
  Assessment 2 (Week 17): number analyzed (Participants) | 129 | 89
  Assessment 2 (Week 17) | 2.74 [0.24 to 5.25] | 5.78 [2.80 to 8.75]
  Assessment 3 (Week 25): number analyzed (Participants) | 101 | 68
  Assessment 3 (Week 25) | 4.58 [1.80 to 7.35] | 7.92 [4.58 to 11.27]
  Assessment 4 (Week 33): number analyzed (Participants) | 74 | 43
  Assessment 4 (Week 33) | 4.08 [0.92 to 7.23] | 5.83 [1.77 to 9.89]
  Assessment 5 (Week 41): number analyzed (Participants) | 53 | 32
  Assessment 5 (Week 41) | 6.73 [3.09 to 10.37] | 5.12 [0.50 to 9.74]
  Assessment 6 (Week 49): number analyzed (Participants) | 37 | 23
  Assessment 6 (Week 49) | 3.91 [-0.35 to 8.16] | 10.85 [5.49 to 16.21]

12. Secondary Outcome: Change From Baseline in the European Quality of Life Five Dimensions Questionnaire (EQ-5D-5L) - Health Utility Index (HUI)
Description: The European Quality of Life 5D-5L Scale (EQ-5D-5L) assesses general health-related quality of life. Health is defined in 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Responses are coded so that a '1' indicates no problem, and '5' indicates the most serious problem. The responses for the 5 dimensions are combined in a 5-digit number. The EQ-5D-5L health utility index (HUI) is assessed using the Crosswalk algorithm for France based on the individual responses to the 5 EQ-5D-5L domains ranging from -0.530 to 1.000. The smallest change considered clinically meaningful, is defined as a score difference of 0.08 points.
Time Frame: Clinic visit closest to the disease evaluation on weeks 9, 17, 25, 33, 41, 49.
Population: Intent-to-Treat population (all randomized participants) with available scores for each assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Nivolumab and Sitravatinib | Docetaxel
Number analyzed (Participants) | 193 | 154
Score on a scale
  Assessment 1 (Week 9) | -0.09 [-0.12 to -0.06] | -0.05 [-0.08 to -0.01]
  Assessment 2 (Week 17): number analyzed (Participants) | 140 | 101
  Assessment 2 (Week 17) | -0.07 [-0.11 to -0.04] | -0.10 [-0.14 to -0.06]
  Assessment 3 (Week 25): number analyzed (Participants) | 108 | 74
  Assessment 3 (Week 25) | -0.10 [-0.14 to -0.06] | -0.15 [-0.20 to -0.10]
  Assessment 4 (Week 33): number analyzed (Participants) | 78 | 46
  Assessment 4 (Week 33) | -0.09 [-0.13 to -0.04] | -0.09 [-0.15 to -0.03]
  Assessment 5 (Week 41): number analyzed (Participants) | 56 | 34
  Assessment 5 (Week 41) | -0.08 [-0.14 to -0.03] | -0.12 [-0.18 to -0.05]
  Assessment 6 (Week 49): number analyzed (Participants) | 42 | 23
  Assessment 6 (Week 49) | -0.10 [-0.16 to -0.04] | -0.15 [-0.23 to -0.07]

13. Secondary Outcome: Change From Baseline in the European Quality of Life Five Dimensions Questionnaire (EQ-5D-5L) - Visual Analogue Score (VAS)
Description: The Visual Analogue Score (VAS) is a component of the EQ-5D-5L and assesses the patient's self-rated health using a vertical visual analogue scale where numbered 0 (the worst health you can image) to 100 (the best health you can imageine). The smallest change considered clinically meaningful, is defined as a score difference of 7 points.
Time Frame: Clinic visit closest to the disease evaluation on weeks 9, 17, 25, 33, 41, 49.
Population: Intent-to-Treat population (all randomized participants) with available scores for each assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Change in score on a scale
Arm/Group | Nivolumab and Sitravatinib | Docetaxel
Number analyzed (Participants) | 193 | 154
Change in score on a scale
  Assessment 1 (Week 9) | -4.74 [-7.21 to -2.27] | -3.77 [-6.52 to -1.01]
  Assessment 2 (Week 17): number analyzed (Participants) | 140 | 101
  Assessment 2 (Week 17) | -3.24 [-6.03 to -0.45] | -5.12 [-8.37 to -1.86]
  Assessment 3 (Week 25): number analyzed (Participants) | 108 | 74
  Assessment 3 (Week 25) | -3.37 [-6.49 to -0.25] | -8.72 [-12.46 to -4.98]
  Assessment 4 (Week 33): number analyzed (Participants) | 78 | 46
  Assessment 4 (Week 33) | -3.41 [-7.00 to 0.19] | -2.71 [-7.30 to 1.88]
  Assessment 5 (Week 41): number analyzed (Participants) | 56 | 34
  Assessment 5 (Week 41) | -3.55 [-7.71 to 0.61] | -2.89 [-8.17 to 2.38]
  Assessment 6 (Week 49): number analyzed (Participants) | 42 | 23
  Assessment 6 (Week 49) | -6.05 [-10.80 to -1.31] | -4.17 [-10.48 to 2.15]

14. Secondary Outcome: Sitravatinib Plasma Concentration by Time Point
Time Frame: 0.5 hours post dose on cycle 1 (day 1) and 5 hours post dose on cycle 1 (day 1 and 15), and pre-dose on cycle 1 (day 15), and cycle 2, 3, and 5 (day 1)
Population: Pharmacokinetic Evaluable Population - all patients who received treatment with sitravatinib and had sufficient concentration-time data to permit calculation for sitravatinib at each time point
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Nivolumab and Sitravatinib: Participants with Advanced Non-Squamous Non-Small Cell Lung Cancer were administered with Nivolumab by intravenous infusion over 30 minutes at 240 milligram (mg) every 2 weeks or at 480 mg every 4 weeks at the discretion of the investigator. Sitravatinib capsules were administered at 100 mg orally, once daily.
Arm/Group | Nivolumab and Sitravatinib
Number analyzed (Participants) | 227
ng/mL
  Cycle 1 Day 1/ 30 mins Post-Dose: number analyzed (Participants) | 162
  Cycle 1 Day 1/ 30 mins Post-Dose | 2.73201 (4.816044)
  Cycle 1 Day 1/ 5 hours Post-Dose | 32.41228 (21.358205)
  Cycle 1 Day 15/ Pre-Dose: number analyzed (Participants) | 177
  Cycle 1 Day 15/ Pre-Dose | 75.72754 (35.261907)
  Cycle 1 Day 15/ 5 hours Post-Dose: number analyzed (Participants) | 180
  Cycle 1 Day 15/ 5 hours Post-Dose | 89.71667 (36.289115)
  Cycle 2 Day 1/ Pre-Dose: number analyzed (Participants) | 145
  Cycle 2 Day 1/ Pre-Dose | 62.20483 (27.055422)
  Cycle 3 Day 1/ Pre-Dose: number analyzed (Participants) | 84
  Cycle 3 Day 1/ Pre-Dose | 51.90238 (19.946633)
  Cycle 5 Day 1/ Pre-Dose: number analyzed (Participants) | 39
  Cycle 5 Day 1/ Pre-Dose | 50.40513 (24.995304)

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from first dose to primary completion (up to approximately 44 months). SAEs and Other AEs were assessed from first dose up to 28 days post last dose, and up to 100 days post last dose of nivolumab for immune-related AEs (Up to maximum of 38 months)
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for SAE and Other (Not Including Serious) AE represents all participants that received at least 1 dose of study medication.
  Adverse event analysis was pre-specified to be assessed per arm and not per dose/ capsule formulation since the nivolumab doses and sitravatinib capsule formulations were considered equivalent and interchangeable for the purposes of this study.
Groups:
- Nivolumab and Sitravatinib: Participants with Advanced Non-Squamous Non-Small Cell Lung Cancer were administered with Nivolumab by intravenous infusion over 30 minutes at 240 milligram (mg) every 2 weeks or at 480 mg every 4 weeks at the discretion of the investigator . Sitravatinib malate capsules were administered at 100 mg orally, once daily (QD).
Arm/Group | Nivolumab and Sitravatinib | Docetaxel
All-Cause Mortality (participants affected / at risk) | 200/284 | 216/293
Serious Adverse Events (participants affected / at risk) | 126/281 | 101/273
Other Adverse Events (participants affected / at risk) | 277/281 | 270/273
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab and Sitravatinib (N=281) | Docetaxel (N=273)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 10 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 16 | 13
Sepsis (Infections and infestations) | 3 | 5
Pneumonia bacterial (Infections and infestations) | 2 | 0
Pneumonia viral (Infections and infestations) | 2 | 2
Urinary tract infection (Infections and infestations) | 2 | 2
Abdominal sepsis (Infections and infestations) | 1 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 1
Coronavirus infection (Infections and infestations) | 1 | 3
Device related infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 3
Gastroenteritis (Infections and infestations) | 1 | 0
Groin abscess (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Periumbilical abscess (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Vestibular neuronitis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 2
COVID-19 (Infections and infestations) | 0 | 2
Colonic abscess (Infections and infestations) | 0 | 2
Escherichia infection (Infections and infestations) | 0 | 1
Infectious pleural effusion (Infections and infestations) | 0 | 1
Pneumonia necrotising (Infections and infestations) | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Tuberculosis (Infections and infestations) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 26 | 6
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Colitis (Gastrointestinal disorders) | 7 | 1
Vomiting (Gastrointestinal disorders) | 5 | 4
Diarrhoea (Gastrointestinal disorders) | 4 | 4
Nausea (Gastrointestinal disorders) | 3 | 4
Intestinal perforation (Gastrointestinal disorders) | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Jejunal perforation (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Neutropenic colitis (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 3 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Immune-mediated myocarditis (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Prinzmetal angina (Cardiac disorders) | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 2
Cardiac failure (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Fluid overload (Cardiac disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 4 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 4 | 1
Ataxia (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 1
Radiculopathy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 5
Toxic encephalopathy (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 3 | 2
Hydronephrosis (Renal and urinary disorders) | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 0
Renal impairment (Renal and urinary disorders) | 2 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Neurogenic bladder (Renal and urinary disorders) | 0 | 1
Fatigue (General disorders) | 2 | 2
Asthenia (General disorders) | 1 | 2
Death (General disorders) | 1 | 1
General physical health deterioration (General disorders) | 1 | 5
Euthanasia (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 2
Coronavirus test positive (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Myocardial necrosis marker increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Blood lactic acid increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 1
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 3 | 0
Hypotension (Vascular disorders) | 2 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Embolism arterial (Vascular disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 13
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Mental status changes (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 2
Vertigo (Ear and labyrinth disorders) | 1 | 0
Glaucoma (Eye disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab and Sitravatinib (N=281) | Docetaxel (N=273)
Diarrhoea (Gastrointestinal disorders) | 178 | 107
Nausea (Gastrointestinal disorders) | 100 | 98
Vomiting (Gastrointestinal disorders) | 74 | 51
Constipation (Gastrointestinal disorders) | 68 | 62
Stomatitis (Gastrointestinal disorders) | 52 | 52
Abdominal pain (Gastrointestinal disorders) | 46 | 22
Dyspepsia (Gastrointestinal disorders) | 29 | 15
Dry Mouth (Gastrointestinal disorders) | 24 | 10
Abdominal Pain Upper (Gastrointestinal disorders) | 18 | 10
Weight decreased (Investigations) | 91 | 32
Alanine aminotransferase increased (Investigations) | 43 | 4
Aspartate aminotransferase increased (Investigations) | 40 | 4
Blood alkaline phosphatase increased (Investigations) | 24 | 7
Lipase increased (Investigations) | 24 | 10
Blood thyroid stimulating hormone increased (Investigations) | 22 | 6
Amylase increased (Investigations) | 21 | 8
Blood creatinine increased (Investigations) | 21 | 6
White blood cell count decreased (Investigations) | 3 | 35
Neutrophil count decreased (Investigations) | 2 | 88
Fatigue (General disorders) | 99 | 113
Asthenia (General disorders) | 53 | 72
Oedema peripheral (General disorders) | 29 | 53
Non-cardiac chest pain (General disorders) | 19 | 8
Pyrexia (General disorders) | 17 | 30
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 62 | 59
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 57 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 55 | 32
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 18 | 8
Productive cough (Respiratory, thoracic and mediastinal disorders) | 18 | 12
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 16 | 4
Decreased appetite (Metabolism and nutrition disorders) | 108 | 82
Hypomagnesaemia (Metabolism and nutrition disorders) | 38 | 34
Dehydration (Metabolism and nutrition disorders) | 23 | 26
Hyponatraemia (Metabolism and nutrition disorders) | 23 | 17
Hypokalaemia (Metabolism and nutrition disorders) | 22 | 19
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 49 | 5
Rash (Skin and subcutaneous tissue disorders) | 32 | 19
Dry skin (Skin and subcutaneous tissue disorders) | 25 | 13
Pruritus (Skin and subcutaneous tissue disorders) | 23 | 13
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 85
Arthralgia (Musculoskeletal and connective tissue disorders) | 43 | 35
Back pain (Musculoskeletal and connective tissue disorders) | 34 | 21
Muscular weakness (Musculoskeletal and connective tissue disorders) | 26 | 20
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20 | 12
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 17 | 16
Muscle spasms (Musculoskeletal and connective tissue disorders) | 15 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 13 | 30
Bone pain (Musculoskeletal and connective tissue disorders) | 12 | 22
Hypertension (Vascular disorders) | 105 | 14
Hypotension (Vascular disorders) | 7 | 24
Coronavirus infection (Infections and infestations) | 27 | 9
Urinary tract infection (Infections and infestations) | 16 | 18
Pneumonia (Infections and infestations) | 14 | 16
Headache (Nervous system disorders) | 33 | 15
Dizziness (Nervous system disorders) | 31 | 20
Dysgeusia (Nervous system disorders) | 28 | 43
Peripheral sensory neuropathy (Nervous system disorders) | 8 | 19
Paraesthesia (Nervous system disorders) | 6 | 26
Neuropathy peripheral (Nervous system disorders) | 4 | 24
Hypothyroidism (Endocrine disorders) | 85 | 6
Fall (Injury, poisoning and procedural complications) | 11 | 16
Insomnia (Psychiatric disorders) | 13 | 26
Anaemia (Blood and lymphatic system disorders) | 21 | 62
Leukopenia (Blood and lymphatic system disorders) | 2 | 19
Neutropenia (Blood and lymphatic system disorders) | 0 | 72
Lacrimation increased (Eye disorders) | 1 | 16

LIMITATIONS AND CAVEATS:
Participants enrolled in the USA who began treatment with the sitravatinib free base capsule formulation prior to protocol amendment 03 will remain on the free base capsule formulation throughout the duration of the study; the starting dose of sitravatinib free base capsule formulation was 120 mg QD.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-07): https://cdn.clinicaltrials.gov/large-docs/71/NCT03906071/Prot_SAP_000.pdf